CLINICAL TRIAL: NCT05291234
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Efficacy, Pharmacokinetics and Pharmacodynamics of ABBV-916 in Subjects With Early Alzheimer's Disease
Brief Title: A Study to Assess Safety of ABBV-916 and How Intravenous ABBV-916 Moves Through Body and Affects Brain Amyloid Plaque Clearance in Adult Participants (Aged 50-90 Years) With Early Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M22-721; 2022-500691-59-00 (Other: EU CT)
Record Dates: First submitted 2022-03-21; First posted 2022-03-22 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer's Disease (AD)
Keywords: Alzheimer's Disease (AD); Early Alzheimer's Disease; ABBV-916
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Stage A: ABBV-916 (Experimental): Participants will receive ABBV-916 for 24 weeks. Participants at the end of 24 weeks will have the option of participating in the 2-year Extension Period.
  Interventions: Drug: ABBV-916
- Stage A: Placebo for ABBV-916 (Placebo Comparator): Participants will receive Placebo for 24 weeks. Participants at the end of 24 weeks will have the option of participating in the 2-year Extension Period.
  Interventions: Drug: Placebo
- Stage B: ABBV-916 Dose A (Experimental): Participants will receive ABBV-916 Dose A for 24 weeks. Participants at the end of 24 weeks will have the option of participating in the 2-year Extension Period.
  Interventions: Drug: ABBV-916
- Stage B: Placebo for ABBV-916 (Placebo Comparator): Participants will receive Placebo for 24 weeks. Participants at the end of 24 weeks will have the option of participating in the 2-year Extension Period.
  Interventions: Drug: Placebo
- Stage B: ABBV-916 Dose B (Experimental): Participants will receive ABBV-916 Dose B for 24 weeks. Participants at the end of 24 weeks will have the option of participating in the 2-year Extension Period.
  Interventions: Drug: ABBV-916

INTERVENTIONS:
Drug: ABBV-916 — Intravenous administration
  Arms: Stage A: ABBV-916; Stage B: ABBV-916 Dose A; Stage B: ABBV-916 Dose B
Drug: Placebo — Intravenous administration
  Arms: Stage A: Placebo for ABBV-916; Stage B: Placebo for ABBV-916

SUMMARY:
Alzheimer's disease (AD) is a progressive, irreversible neurological disorder and is the most common cause of dementia in the elderly population. Clinical symptoms of the disease may begin with occasional forgetfulness such as misplacement of items, forgetting important dates or events, and may progress to noticeable memory loss, increased confusion and agitation, and eventually, loss of independence and non-responsiveness. This study will assess how safe and effective ABBV-916 is in treating early AD. Adverse events, change in disease activity, and how ABBV-916 moves through body of participants will be assessed.

ABBV-916 is an investigational drug being developed for the treatment of early AD. This study is conducted in 2 stages. Stage A is a multiple ascending dose study. There is a 1 in 4 chance that participants are assigned to receive placebo. Stage B is a proof-of-concept study. In Stage B, there is a 1 in 5 chance that participants will be assigned to receive placebo. The first 6 months of this study are "double-blind," which means that neither the trial participant nor the study doctors know which treatments will be given. This will be followed by a 2-year extension period in which all participants will receive ABBV-916. Approximately 195 participants aged 50-90 years will be enrolled in about 90 sites across the world.

Participants will receive intravenous (IV) doses of ABBV-916 or placebo once every 4 weeks (Q4W) for 24 weeks and will be followed for an additional 16 weeks. Participants will have the option of participating in a 2-year, open-label, Extension Period receiving IV ABBV-916.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, magnetic resonance imaging (MRI), blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Stage 3 or Stage 4 Alzheimer's disease (AD) based on the 2018 National Institute on Aging (NIA)-Alzheimer's Association (AA) Research Framework Criteria.

  * Mini-Mental State Examination (MMSE) score of 20 to 28, inclusive, at Screening.
  * Blood-based biomarker results with a value consistent with amyloid positron emission tomography (PET) positivity. The biomarker will be chosen by the sponsor and described in the Laboratory Manual. Biomarker results will not be required for eligibility if the participant has a positive Amyloid PET scan meeting the central reader criteria.
* Amyloid PET scan results consistent with amyloid pathology.
* Stage B: Participants must have a study partner who spends a minimum average of 10 hours per week with the participant.

Exclusion Criteria:

* Significant pathological findings on brain MRI at screening including, but not limited to, evidence of vasogenic edema, 4 or more microhemorrhages, any macrohemorrhages, any superficial siderosis, or severe white matter disease.
* Any anticoagulants or have a bleeding disorder that is not adequately controlled.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2025-11-19 (Actual); Study Completion 2025-11-19 (Actual)

PRIMARY OUTCOMES:
Number of Participants Experiencing Adverse Events (AEs) | Up to approximately 160 weeks
  An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study.
Stage A: Maximum Observed Serum Concentration (Cmax) for Multiple Ascending Dose of ABBV-916 | Up to approximately 24 weeks
  Cmax of ABBV-916 will be determined.
Stage A: Time to Cmax (Tmax) for Multiple Ascending Dose of ABBV-916 | Up to approximately 24 weeks
  Tmax of ABBV-916 will be determined.
Stage A: Apparent Terminal Phase Elimination Rate Constant (β) of ABBV-916 | Up to approximately 24 weeks
  Apparent terminal phase elimination rate constant (β) of ABBV-916 will be determined.
Stage A: Terminal Phase Elimination Half-Life (t1/2) of ABBV-916 | Up to approximately 24 weeks
  T1/2 of ABBV-916 will be determined.
Stage A: Trough Serum Concentration (Ctrough) of ABBV-916 at the End of a Dosing Interval | Up to approximately 24 weeks
  Ctrough of ABBV-916 will be determined.
Stage A: Area Under the Concentration-Time Curve (AUC) of ABBV-916 | Up to approximately 24 weeks
  AUC of ABBV-916 will be determined.
Stage A: Cerebrospinal Fluid (CSF) Concentration as a Measure of ABBV-916 Crossing the Blood Brain Barrier | Up to approximately 24 weeks
  The central value for ratio of ABBV-916 concentration in cerebrospinal fluid (CSF) to that in serum will be estimated for evaluation of the fraction of ABBV-916 crossing the blood brain barrier.
Stage A: Percentage of Participants With Antidrug Antibodies (ADA) as a Measure of Immunogenicity Following Multiple Ascending Dose of ABBV-916 | Up to approximately 24 weeks
  Antidrug antibody (ADA) classification and titers for positive ADA samples will be determined.
Stage B: Change in Brain Amyloid Plaque Deposition (Amyloid Centiloid Value) | Baseline (Week 0) through Week 24
  Change from baseline in brain amyloid plaque deposition (amyloid centiloid value) is measured by amyloid positron emission tomography (PET) scan.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (32):
- United States (32):
  - Tucson Neuroscience Research /ID# 244957, Tucson, Arizona
  - Irvine Clinical Research /ID# 239469, Irvine, California
  - Artemis Institute for Clinical Research - San Diego /ID# 244508, San Diego, California
  - Pacific Research Network, Inc. /ID# 244083, San Diego, California
  - Syrentis Clinical Research /ID# 239682, Santa Ana, California
  - Aventura Neurological Associates /ID# 243892, Aventura, Florida
  - Charter Research - Lady Lake /ID# 244657, Lady Lake, Florida
  - JEM Research Institute /ID# 239122, Lake Worth, Florida
  - ClinCloud - Maitland /ID# 244507, Maitland, Florida
  - ClinCloud LLC - Viera/Melbourne /ID# 240635, Melbourne, Florida
  - Merritt Island Medical Research /ID# 239495, Merritt Island, Florida
  - Optimus U /ID# 245868, Miami, Florida
  - Finlay Medical Research /ID# 245996, Miami, Florida
  - Allied Biomedical Res Inst Inc /ID# 244823, Miami, Florida
  - Renstar Medical Research /ID# 240153, Ocala, Florida
  - K2 Medical Research - Ocoee /ID# 246849, Ocoee, Florida
  - K2 Medical Research - Orlando - South Orlando Avenue /ID# 243919, Orlando, Florida
  - Charter Research - Winter Park /ID# 244778, Orlando, Florida
  - Headlands Research - Orlando /ID# 239119, Orlando, Florida
  - Neurology Associates Ormond Beach /ID# 245527, Ormond Beach, Florida
  - IMIC Inc. Medical Research /ID# 245900, Palmetto Bay, Florida
  - Alzheimer's Research and Treatment Center - Stuart /ID# 245477, Stuart, Florida
  - Alzheimer's Research and Treatment Center - Wellington /ID# 245201, Wellington, Florida
  - Premiere Research Institute - Palm Beach /ID# 240108, West Palm Beach, Florida
  - Clinical Site Partners (CSP) - Orlando /ID# 245127, Winter Park, Florida
  - Conquest Research /ID# 243916, Winter Park, Florida
  - Columbus Memory Center /ID# 245054, Columbus, Georgia
  - QUEST Research Institute /ID# 239459, Farmington Hills, Michigan
  - Advanced Memory Research Institute of NJ /ID# 239533, Toms River, New Jersey
  - Keystone Clinical Studies LLC /ID# 239973, Plymouth Meeting, Pennsylvania
  - Clinical Trials of Texas, Inc /ID# 244917, San Antonio, Texas
  - Re:Cognition Health - Fairfax VA /ID# 239501, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M22-721